CLINICAL TRIAL: NCT05585476
Title: Effectiveness of C02 Microfractionated Laser in Conjunction With Topical Regenerative Therapy in the Management of Vulvo-vaginal Atrophy in Patients With a History of Breast Cancer. Randomized Experimental and Comparative Study.
Brief Title: A Laser and Topical Treatment Combination in the Vulvo-vaginal Atrophy Management in Breast Cancer Patients.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Investigación Sanitaria de la Fundación Jiménez Díaz (Other)
Collaborators: Lumenis Be Ltd. (Industry); Mucosa Innovations, S.L. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FJD-LCO2-19-01
Record Dates: First submitted 2022-09-21; First posted 2022-10-18 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Female Urogenital Diseases; Breast Cancer Female
Keywords: Vulvovaginal atrophy; Breast cancer; Hormone therapy; Regenerative topical treatment; C02 microfractionated laser
MeSH Terms: conditions — Female Urogenital Diseases; Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: A single-blind, randomized, controlled clinical trial is proposed, in which the patients included will be assigned to one of the three treatment arms.
Who Masked: Participant, Outcomes Assessor
Masking Description: In order to mask the patients from the treatment group to which they have been assigned, a simulated laser treatment session will be carried out in the case of patients belonging to the topical regenerative treatment group, which will consist of keeping the device turned off during it but faithfully reproducing both the duration as the sounds emitted by the device through recording previously made. In the case of patients assigned to laser treatment exclusively, they will be provided with a topical placebo (water-based), which must be applied with the same regimen as the emollient treatment under study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Laser + Regenerative topical treatment (Experimental): The treatments used in this arm are the following:
  1. º Microfractionated laser treatment of C02, through the AcupulseDuo generator of the company Lumenis®. The treatment regimen would consist of three sessions in total with periodicity of 4 weeks, between the first and the second, and 6 weeks between the second and third. The application of laser energy will be carried out by vaginal and vulvar terminals. The dose applied will consist of monopulse shots distributed throughout the vaginal mucosa and vulvar skin of 10 mJ of energy and at a density of 10%.
  2. nd Topical treatment: It consists of the application of XCM® intim of the company Mucosa Innovations. The route of administration would be vulvo-vaginal. The dose applied would be 2 ml of total product every 12 hours during 36 months.
  Interventions: Device: C02 microablative laser; Combination Product: Regenerative topical treatment
- Regenerative topical treatment (Experimental): In this arm, only the regenerative treatment of XCM® intim of the company Mucosa Innovations will be used. The route of administration would be vulvo-vaginal. The dose applied would be 2 ml of total product every 12 hours. The total duration of treatment would be 36 months.
  Interventions: Combination Product: Regenerative topical treatment
- Laser treatment (Experimental): The treatments used in this arm are the following:
  1. º Microfractionated laser treatment of C02, through the AcupulseDuo generator of the company Lumenis®. The treatment regimen would consist of three sessions in total with periodicity of 4 weeks, between the first and the second, and 6 weeks between the second and third. The application of laser energy will be carried out by vaginal and vulvar terminals. The dose applied will consist of monopulse shots distributed throughout the vaginal mucosa and vulvar skin of 10 mJ of energy and at a density of 10%.
  2. ºPlacebo vulvo-vaginal topical gel, consisting of a watery base.
  Interventions: Device: C02 microablative laser

INTERVENTIONS:
Device: C02 microablative laser — The C02 microablative laser was the first to be used in the treatment of menopausal genitourinary syndrome. Its mechanism of action is based on the emission of light at a wavelength of 10600nm that is absorbed by the water molecules contained in the vaginal mucosa, leading to local remodeling of connective tissue and neoformation of collagen, elastic fibers and other components of the extracellular matrix.
  Arms: Laser + Regenerative topical treatment; Laser treatment
Combination Product: Regenerative topical treatment — It is a moisturizing and regenerating gel whose active ingredients are olive oil, trimethylglycine and xylitol.
  Arms: Laser + Regenerative topical treatment; Regenerative topical treatment

SUMMARY:
The genito-urinary syndrome of menopause severely affects patients with a history of gynecological cancer, especially those diagnosed with breast cancer. At the present time, we do not have solid scientific evidence on treatments that can be effective and safe to address this pathology. Based on the above, we have developed our working hypothesis where it is postulated that the microfractionated laser treatment of C02, in conjunction with topical regenerative treatment, constitute an effective alternative in the management of vulvo-vaginal atrophy in oncological patients who have contraindicated hormonal treatments.

DETAILED DESCRIPTION:
Based on the hypothesis set out in the previous section, the main objective of the study will consist of:

-To assess the effectiveness of microfractionated C02 laser therapy in combination with non-hormonal topical regenerative therapy versus laser treatment or non-hormonal topical regenerative treatment (the latter two exclusively) in the management of symptoms derived from vulvovaginal atrophy in cancer patients who are contraindicated to the use of hormonal therapies.

As secondary objectives we have the following:

* To determine the prevalence and incidence of genitourinary syndrome in our population of patients diagnosed with breast cancer and who are undergoing adjuvant or neoadjuvant treatment (with the exception of chemotherapy).
* To assess the impact of genitourinary syndrome on the quality of life of these patients.
* To determine the degree of correlation between intensity of the symptomatology and impact on the quality of life of the same with the presence of characteristic changes of hormonal depletion at the tissue level and vaginal microbiota.
* To evaluate the safety and tolerability of the C02 laser in our group of patients. Special attention will be paid to the occurrence of adverse events that have not been described in the literature at the present time.
* Describe other effects of laser treatment on urinary symptoms that could serve as hypotheses for future studies.
* To evaluate the safety and tolerability of the topical non-hormonal regenerating agent XCM intim in our group of patients.
* To describe the effects of topical non-hormonal regenerative therapy on vulvo-vaginal and urinary symptoms and the impact on the quality of life of these patients.

To carry out all the above, it is proposed to perform a controlled and randomized clinical trial, single blind, in which the patients included will be assigned to one of the 3 existing treatment arms and that we will explain in detail in later sections.

Recruitment is planned to begin in December 2022. The overall duration of the study is estimated at approximately 42 months, from the beginning of the recruitment period to the last follow-up visit. This study is intended to be conducted from December 2022 to January 2026.

All those patients who meet the inclusion criteria and do not present any reason for exclusion will be given the informative document on the study. If they agree to participate, they will deliver said signed document and will be recruited and randomized in a single-blind manner (only the participant), in a 1:1:1 ratio to laser treatment + regenerative topical treatment or to regenerative topical treatment or to laser treatment ( latter 2 in exclusivity). The entire process of selection, inclusion and randomization will be supervised by both the Research Institute and the Clinical Research Ethics Committee of the Jiménez Díaz Foundation, which will carry out regular audits.

The study will be conducted in accordance with the protocol and standards of good clinical practice, as described in: Harmonized Tripartite Standards of ICH E6, for Good Clinical Practice 1996. Law 14/2007 on Biomedical Research Directive 2001/20/EC. Updated Declaration of Helsinki and amendments concerning medical research on human beings. The researcher agrees, with the signing of this protocol, to follow the instructions and procedures described therein and therefore will comply with the principles of Good Clinical Practice on which it is based. Once the protocol has been signed, it should not be modified without the written agreement of both the sponsor and the principal investigator, and with the consent of the Clinical Trials Ethics Committee.

All the information collected will be treated in a strictly confidential manner, in accordance with current regulations (Regulation (EU) 2016/679 of the European Parliament and of the Council, of April 27, 2016 (GDPR), Law 41/2002 on Patient Autonomy, Law 14/1986 General Health and Law 14/2007 on Biomedical Research). The patient will have the right to access, modify, oppose and cancel their data. In addition, they can limit the processing of data that are incorrect, request a copy or transfer to a third party (portability) the data that has been provided for the study. To exercise their rights, the patient must contact the principal investigator of the study. Data cannot be deleted even if the patient stops participating in the trial to ensure the validity of the research and comply with legal duties and drug authorization requirements. Likewise, the patient has the right to contact the Data Protection Agency if they are not satisfied.

It is the investigator's responsibility to document all adverse events that occur during the clinical trial. At each visit/assessment, all adverse events observed by both the investigator and one of his or her clinical collaborators, as well as those reported by the subject spontaneously or in response to a direct question, shall be evaluated by the investigator and noted in the adverse events section of the subject's data collection notebook.

The nature of each event, the time of onset after the intervention, the duration, the severity and relationship to the intervention should be established. The details of its handling must be recorded on the corresponding pages of the data collection notebook. The initial symptomatology should be well documented at the screening visit. It is important to correctly collect the baseline information in order to interpret the data of the following visits.

Investigators should follow up on subjects with adverse events until they have subsided, disappeared, or until the process has stabilized. Reports on the course of the subject's evolution should be sent to the monitor of the clinical trial.

The principal investigator shall report serious and unexpected adverse events to the sponsor by telephone or fax within 24 hours of becoming aware of the adverse event by the investigator, who shall in turn inform the health authorities. The previous report made by telephone or fax shall be followed by a complete report including a copy of the relevant data collected or recorded at the centre or other documents that occur as a result of the adverse event.

The total number of visits for patients in both treatment arms will be 8, leaving the study schedule as follows:

* Consult before treatment.
* First treatment visit (after acceptance and signing of the informed consent): First session of laser treatment and initiation of topical treatment.
* Second treatment visit (one month after the first session): Second session of laser treatment and topical treatment control.
* Third treatment visit (6 weeks after the second session): Third session of laser treatment and topical treatment control.
* Review 1.5 months after the 3rd session.
* Review 6 months after the 3rd session.
* Review 12 months after the 3rd session.
* Review 24 months after the 3rd session.

The tests and studies to be carried out during the study will be the following:

* Anamnesis (in all visits).
* Physical examination (at all visits).
* Gynecological ultrasound (in 1st visit, before starting treatment).
* Validated questionnaires (in all visits).
* Measurements of skin characteristics with cutometer (at all visits).
* Vaginal exudate (in first pretreatment visit, visit of the month and a half of finishing laser treatment, visit of the 6 months after finishing the laser treatment session, visit of the 12 months and visit of the 24 months).
* Vaginal mucosal biopsy (at the 1st visit before starting treatment and a month and a half after the third session).

A digital data collection notebook will be created by the company Xolomon ® to guarantee the quality and reliability of the information. All data will be entered 2 times by 2 different researchers between whom there will be no contact. In the event that there is a discrepancy in the same field, the computer system will send an alert to the main researcher and he will be in charge of clarifying where the error is. Likewise, it will be the principal investigator who verifies the integrity, accuracy and veracity of the data entered, by comparing them with those collected in the clinical history of patient care.

All variables entered in the digital data notebook will have masks, ranges of values and dictionaries depending on the type of variable and the content they must integrate.

Regarding the statistical analysis of the data, a description of the characteristics of the patients will be made. Qualitative variables will be described by frequencies and percentages. The quantitative variables will be described by the mean and the standard deviation, or by the median and the interquartile range, depending on the degree of symmetry presented by the distribution of the data. Comparisons between the two treatment groups referring to the qualitative variables will be made by the Chi-square test, or failing that by Fisher's exact test. In the case of quantitative variables, comparisons will be made by Student's t test, or by Wilcoxon range test, depending on whether or not the data follow a normal distribution. To test normality, the Shapiro-Wilk test will be used. Whenever possible, the difference between the two treatment groups will be quantified, along with their 95% confidence intervals. The treatment of the lost values will be carried out through the Multiple Imputation method, for which, sets of databases will be generated from the original database, which will contain imputed values based on a random selection. The statistical analyses will be carried out by the Biostatistics service of the Jiménez Díaz Foundation University Hospital, through the Statistical Program Stata 14.0.

The sample size has been calculated in order to detect a difference of 2 points, between the means of the symptom intensity scale of the three groups. A maximum standard deviation of 3 points and a loss percentage of 10% are assumed. Under these assumptions, if we set the significance level at 5% and statistical power at 90%, 60 patients in each group would be

ELIGIBILITY:
Inclusion Criteria:

Patients must meet ALL of the following criteria to be included in the study:

1. Patients over 18 years of age
2. Who have a history of breast malignancy, and are on adjuvant or neoadjuvant treatment with hormone therapy.
3. That they suffer symptoms related to vulvo-vaginal atrophy and thus become evident to the gynecological examination (Vaginal Health Index<ó=15).
4. That this clinic significantly affects your quality of life ( score in Sexual Function-Vaginal Changes Questionnaire less than or equal to 24 points).
5. Who have not received any treatment for vulvo-vaginal atrophy in at least the previous 6 months. Purely moisturizing or emollient treatments that do not contain any regenerating substance (hyaluronic acid, gotu kola, vitamin E or rosehip oil) are not considered exclusive.
6. That they agree to participate and give their written I consent.

Exclusion Criteria:

Patients who present ANY of the following criteria may not be selected to participate in this study:

1. Medical or surgical history that at the discretion of the researcher does not allow participation in the study.
2. Refusal to participate in the study and to sign consent.
3. Be on chemotherapy treatment at the time of inclusion in the study.
4. Have completely completed the adjuvant hormonal treatment.
5. Have a history of vulvar, vaginal and/or cervical malignancy.
6. Have received radiation therapy to the pelvic and/or genital region.
7. Sjögren's syndrome and other pathologies that occur with mucosal involvement.
8. Present any type of disease that occurs with alteration of collagenogenesis.
9. Intake of other cytotoxic drugs that lead to mucositis and alterations of tissue regeneration in the last 6 months.
10. Have previously received laser and/or radiofrequency treatment for the treatment of genital atrophy or other pelvic floor dysfunctions.
11. Active urinary and/or genital tract infection.
12. Diagnosis of gestation at the time of recruitment.
13. History of malignant neoplasm of the urinary tract.
14. Have severe stress urinary incontinence (Sandvik test with a score equal to or greater than 8)
15. Diagnosis of pelvic organ prolapse grade III or higher according to the POP-Q classification.
16. Any other condition which, in the opinion of the investigator, means that the patient is not in a position to understand the implication of participating in the study and/or of following the established procedures.

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Presence of symptoms at the vulvovaginal level and their intensity | From prior consultation at the beginning of treatment to 24 months after it ends.
  This group will include the following items:
  * Pain with sexual intercourse (dyspareunia).
  * Feeling of vaginal stiffness.
  * Dryness.
  * Vulvar itching.
  * Vulvar and/or vaginal burning.
  * Urinary frequency (more than 8 times a day).
  * Burning when urinating (dysuria). The way to measure the intensity of these symptoms will be through Visual Analog Scale Of Symptom Intensity, with absolute values ranging from 0 to 10.
  We will consider improvement a reduction of 2 or more points in at least 50% of the items. Meeting only this item is already considered an efficacy criterion.
Impact in the quality of life of vulvo-vaginal symptoms. | From prior consultation at the beginning of treatment to 24 months after it ends.
  The tool used will be the Sexual Function-Vaginal Changes Questionnaire. Scores equal to or less than 24 points will result in an impact on quality of life. A rise of 3 or more points is considered a significant improvement.
  The severity levels of quality of life impairment will be as follows:
  * Mild (scores between 24 and 17)
  * Moderate (scores between 16 and 8)
  * Severe (scores between 7 and 1)
Changes in vulvar physical examination | From prior consultation at the beginning of treatment to 24 months after it ends.
  We will use the following measurement system:
  Vulvar Health Index Score. It is based on the macroscopic inspection of the vulva performed through a colposcope. The scores range from 0 to 24, being higher to greater atrophy. It is considered a diagnosis of atrophy scores greater than 8 or having obtained 3 points in any of the items. The degrees of gravity are set as follows:
  1. Between 9 and 14 points, mild
  2. Between 15 and 20 points, moderate
  3. Between 21 and 24 points, severe.
  A reduction of 3 or more points in the overall score or at least one point will be considered a favorable response if there has been an item with a score of 3.
Changes in vaginal physical examination | From prior consultation at the beginning of treatment to 24 months after it ends.
  We will use the following measurement systems:
  Vaginal Health Index Score. It is based on the macroscopic inspection of the vagina performed through a colposcope. Scores range from 5 to 25 points (scores equal to or less than 15 are considered diagnostic of atrophy). It is carried out by assessing different items related to exploratory findings.
  We can categorize the scores into different degrees of severity of vulvo-vaginal atrophy objectified to the examination:
  1. >from 15 points, absence of atrophy
  2. Between 15 and 13 points, mild
  3. Between 12 and 9 points, moderate
  4. Between 8 and 5 points, severe
  An increase of 2 or more points in the overall score will be considered a favourable response.
Thickness of the vaginal epithelium | From prior consultation at the beginning of treatment to 24 months after it ends.
  The collection of the sample will consist of taking biopsy of vaginal mucosa using a 4 mm punch as an instrument.
  Once obtained, the sample will be stained with hematoxylin-eosin and subjected to microscopic assessment.
  The unit of measurement shall be in nanometers.
Quantification of cellular glycogen | From prior consultation at the beginning of treatment to 24 months after it ends.
  The collection of the samples will consist of taking biopsies of vaginal mucosa using a 4 mm punch as an instrument.
  The sample will undergo the Schiff technique (PAS) and the number of stained cells will be determined.
Number of capillaries in vaginal mucosa | From prior consultation at the beginning of treatment to 24 months after it ends.
  The collection of samples will consist of taking biopsies of vaginal mucosa using a 4 mm punch as an instrument.
  The immunohistochemical technique will be applied with antibodies against CD31 and a quantitative assessment of the number of capillaries / field of 40 increases will be carried out.
Amount of Lactobacillus in vaginal microbiota | From prior consultation at the beginning of treatment to 24 months after it ends.
  It will be measured through microbiological study. Samples shall be obtained by vaginal exudate.
  The measurements will be made by WERFEN system and PCR technique.
Amount of Candida spp in vaginal microbiota | From prior consultation at the beginning of treatment to 24 months after it ends.
  It will be measured through microbiological study. Samples shall be obtained by vaginal exudate.
  The measurements will be made by WERFEN system and PCR technique.
Amount of Gardnerella vaginalis in vaginal microbiota | From prior consultation at the beginning of treatment to 24 months after it ends.
  It will be measured through microbiological study. Samples shall be obtained by vaginal exudate.
  The measurements will be made by WERFEN system and PCR technique.
Free glycogen detection in vaginal discharge | From prior consultation at the beginning of treatment to 24 months after it ends.
  It will be measured through microbiological study. Samples shall be obtained by vaginal exudate.
  Free glycogen detection will be performed using a commercial kit.
Vaginal pH | From prior consultation at the beginning of treatment to 24 months after it ends.
  It will be measured through microbiological study. Samples shall be obtained by vaginal exudate.
Skin elasticity | From prior consultation at the beginning of treatment to 24 months after it ends.
  It will be performed with the Dual cutometer MPA 580 ® and will determine different characteristics of the vulvar skin.
  The value will be given in the unit of measurement N / m².
Amount of transdermal water in the skin | From prior consultation at the beginning of treatment to 24 months after it ends.
  It will be performed with the Dual cutometer MPA 580 ® and will determine different characteristics of the vulvar skin.
  The value will be given in the unit of measurement g/h/m².
Skin pigmentation | From prior consultation at the beginning of treatment to 24 months after it ends.
  It will be performed with the Dual cutometer MPA 580 ® and will determine different characteristics of the vulvar skin.
  The degree of pigmentation of the skin will be determined based on the concentration of melanin.
Degree of vascularization of the skin | From prior consultation at the beginning of treatment to 24 months after it ends.
  It will be performed with the Dual cutometer MPA 580 ® and will determine different characteristics of the vulvar skin.
  To determine the degree of vascularization of the skin, specific wavelengths will be used, corresponding to the maximum level of spectral absorption of hemoglobin and avoiding other color influences (for example, bilirubin). The result corresponding will be immediately displayed in the form of index figures, on a scale of 0 - 999.

SECONDARY OUTCOMES:
Presence of bladder hyperactivity clinic | From prior consultation at the beginning of treatment to 24 months after it ends.
  The following questionnaires will be used:
  Bladder control self-assessment questionnaire.
  This scale measures 2 items: Presence of symptoms and discomfort generated by them.
  The range of values for each of them goes from 0 to 12, with the severity levels being the following in both cases:
  0-->Absence of symptoms/discomfort. 1-3-->Mild symptoms/discomfort. 4-6-->Moderate symptoms/discomfort. 7-9-->Severe symptoms/discomfort. 10-12-->Very serious symptoms/discomfort.
Presence of urge urinary incontinence | From prior consultation at the beginning of treatment to 24 months after it ends.
  The Sandvik Test will be used. It consists of 2 sections whose scores are multiplied. The range of scores goes from 0 to 12, with the only possible values being 0, 1, 2, 3, 4, 6, 8, 9 and 12. The degree of urinary incontinence shall be classified as follows:
  0-->Absence of incontinence 1-2-->Mild urinary incontinence 3-6-->Moderate urinary incontinence 8-9-->Severe urinary incontinence 12-->Very severe urinary incontinence
Impact of urinary incontinence on quality of life | From prior consultation at the beginning of treatment to 24 months after it ends.
  We will use the International Consultation on Incontinence Questionnaire-Short Form.
  Of this scale we will only use in section that measures the degree of discomfort caused by incontinence and that reaches the values of 1 to 10.

CONTACTS AND LOCATIONS:
Overall Officials: Amalia Cañadas Molina, Principal Investigator — Employee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nappi RE, Particco M, Biglia N, Cagnacci A, Di Carlo C, Luisi S, Paoletti AM. Attitudes and perceptions towards vulvar and vaginal atrophy in Italian post-menopausal women: Evidence from the European REVIVE survey. Maturitas. 2016 Sep;91:74-80. doi: 10.1016/j.maturitas.2016.06.009. Epub 2016 Jun 11. PMID 27451324
- [Background] Amori P, Di Nardo V, Vitiello G, Franca K, Hercogova J, Wollina U, Daaboul F, Tchernev G, Lotti T. Primavera: A new therapeutical approach to vulvo-vaginal atrophy. Dermatol Ther. 2018 Nov;31(6):e12678. doi: 10.1111/dth.12678. Epub 2018 Nov 8. PMID 30411455
- [Background] Palma F, Xholli A, Cagnacci A; as the writing group of the AGATA study. The most bothersome symptom of vaginal atrophy: Evidence from the observational AGATA study. Maturitas. 2018 Feb;108:18-23. doi: 10.1016/j.maturitas.2017.11.007. Epub 2017 Nov 10. PMID 29290210
- [Background] Gandhi J, Chen A, Dagur G, Suh Y, Smith N, Cali B, Khan SA. Genitourinary syndrome of menopause: an overview of clinical manifestations, pathophysiology, etiology, evaluation, and management. Am J Obstet Gynecol. 2016 Dec;215(6):704-711. doi: 10.1016/j.ajog.2016.07.045. Epub 2016 Jul 26. PMID 27472999
- [Background] Mocan-Hognogi RF, Costin N, Malutan A, Ciortea R, Trif IA, Nagy AL, Bogdan ML, Mihu D. Histological changes in the vulva and vagina from ovariectomised rats undergoing oestrogen treatment. Folia Morphol (Warsz). 2016;75(4):467-473. doi: 10.5603/FM.a2016.0026. Epub 2016 Nov 10. PMID 27830882
- [Background] Rozenberg S, Joris A, Albert V, Antoine C, Vandromme J. [La menopause et le traitement hormonal de la menopause : une actualisation]. Rev Med Brux. 2018;39(4):259-263. French. PMID 30320986
- [Background] Sadovsky R, Basson R, Krychman M, Morales AM, Schover L, Wang R, Incrocci L. Cancer and sexual problems. J Sex Med. 2010 Jan;7(1 Pt 2):349-73. doi: 10.1111/j.1743-6109.2009.01620.x. PMID 20092444
- [Background] Trinkaus M, Chin S, Wolfman W, Simmons C, Clemons M. Should urogenital atrophy in breast cancer survivors be treated with topical estrogens? Oncologist. 2008 Mar;13(3):222-31. doi: 10.1634/theoncologist.2007-0234. PMID 18378532
- [Background] Sturdee DW, Panay N; International Menopause Society Writing Group. Recommendations for the management of postmenopausal vaginal atrophy. Climacteric. 2010 Dec;13(6):509-22. doi: 10.3109/13697137.2010.522875. Epub 2010 Sep 30. PMID 20883118
- [Background] Pfeiler G, Glatz C, Konigsberg R, Geisendorfer T, Fink-Retter A, Kubista E, Singer CF, Seifert M. Vaginal estriol to overcome side-effects of aromatase inhibitors in breast cancer patients. Climacteric. 2011 Jun;14(3):339-44. doi: 10.3109/13697137.2010.529967. Epub 2011 Jan 13. PMID 21226657
- [Background] Nappi RE, Palacios S, Particco M, Panay N. The REVIVE (REal Women's VIews of Treatment Options for Menopausal Vaginal ChangEs) survey in Europe: Country-specific comparisons of postmenopausal women's perceptions, experiences and needs. Maturitas. 2016 Sep;91:81-90. doi: 10.1016/j.maturitas.2016.06.010. Epub 2016 Jun 15. PMID 27451325
- [Background] Palacios S, Castelo-Branco C, Currie H, Mijatovic V, Nappi RE, Simon J, Rees M. Update on management of genitourinary syndrome of menopause: A practical guide. Maturitas. 2015 Nov;82(3):308-13. doi: 10.1016/j.maturitas.2015.07.020. Epub 2015 Jul 26. PMID 26261035
- [Background] Tadir Y, Gaspar A, Lev-Sagie A, Alexiades M, Alinsod R, Bader A, Calligaro A, Elias JA, Gambaciani M, Gaviria JE, Iglesia CB, Selih-Martinec K, Mwesigwa PL, Ogrinc UB, Salvatore S, Scollo P, Zerbinati N, Nelson JS. Light and energy based therapeutics for genitourinary syndrome of menopause: Consensus and controversies. Lasers Surg Med. 2017 Feb;49(2):137-159. doi: 10.1002/lsm.22637. Epub 2017 Feb 21. PMID 28220946
- [Background] Gambacciani M, Cervigni M. Erbium laser in gynecology: aims, aspirations and action points. Climacteric. 2015;18 Suppl 1:2-3. doi: 10.3109/13697137.2015.1082258. No abstract available. PMID 26366792
- [Background] Vizintin Z, Lukac M, Kazic M, Tettamanti M. Erbium laser in gynecology. Climacteric. 2015;18 Suppl 1:4-8. doi: 10.3109/13697137.2015.1078668. PMID 26366793
- [Background] Salvatore S, Nappi RE, Zerbinati N, Calligaro A, Ferrero S, Origoni M, Candiani M, Leone Roberti Maggiore U. A 12-week treatment with fractional CO2 laser for vulvovaginal atrophy: a pilot study. Climacteric. 2014 Aug;17(4):363-9. doi: 10.3109/13697137.2014.899347. Epub 2014 Jun 5. PMID 24605832
- [Background] Sokol ER, Karram MM. Use of a novel fractional CO2 laser for the treatment of genitourinary syndrome of menopause: 1-year outcomes. Menopause. 2017 Jul;24(7):810-814. doi: 10.1097/GME.0000000000000839. PMID 28169913
- [Background] Siliquini GP, Tuninetti V, Bounous VE, Bert F, Biglia N. Fractional CO2 laser therapy: a new challenge for vulvovaginal atrophy in postmenopausal women. Climacteric. 2017 Aug;20(4):379-384. doi: 10.1080/13697137.2017.1319815. Epub 2017 May 15. PMID 28503946
- [Background] Gaspar A, Brandi H, Gomez V, Luque D. Efficacy of Erbium:YAG laser treatment compared to topical estriol treatment for symptoms of genitourinary syndrome of menopause. Lasers Surg Med. 2017 Feb;49(2):160-168. doi: 10.1002/lsm.22569. Epub 2016 Aug 22. PMID 27546524
- [Background] Antonino P, Gloria C. A new approach to treatment of vulvo-vaginal atrophy. Maturitas. 2015 Aug;81(4):499. doi: 10.1016/j.maturitas.2015.03.003. Epub 2015 Mar 11. No abstract available. PMID 25835752
- [Background] Filippini M, Del Duca E, Negosanti F, Bonciani D, Negosanti L, Sannino M, Cannarozzo G, Nistico SP. Fractional CO2 Laser: From Skin Rejuvenation to Vulvo-Vaginal Reshaping. Photomed Laser Surg. 2017 Mar;35(3):171-175. doi: 10.1089/pho.2016.4173. Epub 2016 Dec 30. PMID 28056209
- [Background] Murina F, Karram M, Salvatore S, Felice R. Fractional CO2 Laser Treatment of the Vestibule for Patients with Vestibulodynia and Genitourinary Syndrome of Menopause: A Pilot Study. J Sex Med. 2016 Dec;13(12):1915-1917. doi: 10.1016/j.jsxm.2016.10.006. Epub 2016 Nov 15. PMID 27864031
- [Background] Hutchinson-Colas J, Segal S. Genitourinary syndrome of menopause and the use of laser therapy. Maturitas. 2015 Dec;82(4):342-5. doi: 10.1016/j.maturitas.2015.08.001. Epub 2015 Aug 12. PMID 26323234
- [Background] Rabley A, O'Shea T, Terry R, Byun S, Louis Moy M. Laser Therapy for Genitourinary Syndrome of Menopause. Curr Urol Rep. 2018 Aug 17;19(10):83. doi: 10.1007/s11934-018-0831-y. PMID 30117032
- [Background] Salvatore S, Nappi RE, Parma M, Chionna R, Lagona F, Zerbinati N, Ferrero S, Origoni M, Candiani M, Leone Roberti Maggiore U. Sexual function after fractional microablative CO(2) laser in women with vulvovaginal atrophy. Climacteric. 2015 Apr;18(2):219-25. doi: 10.3109/13697137.2014.975197. Epub 2014 Dec 16. PMID 25333211
- [Background] Sokol ER, Karram MM. An assessment of the safety and efficacy of a fractional CO2 laser system for the treatment of vulvovaginal atrophy. Menopause. 2016 Oct;23(10):1102-7. doi: 10.1097/GME.0000000000000700. PMID 27404032
- [Background] Behnia-Willison F, Sarraf S, Miller J, Mohamadi B, Care AS, Lam A, Willison N, Behnia L, Salvatore S. Safety and long-term efficacy of fractional CO2 laser treatment in women suffering from genitourinary syndrome of menopause. Eur J Obstet Gynecol Reprod Biol. 2017 Jun;213:39-44. doi: 10.1016/j.ejogrb.2017.03.036. Epub 2017 Apr 2. PMID 28419911
- [Background] Perino A, Calligaro A, Forlani F, Tiberio C, Cucinella G, Svelato A, Saitta S, Calagna G. Vulvo-vaginal atrophy: a new treatment modality using thermo-ablative fractional CO2 laser. Maturitas. 2015 Mar;80(3):296-301. doi: 10.1016/j.maturitas.2014.12.006. Epub 2014 Dec 25. PMID 25596815
- [Background] Perino A, Cucinella G, Gugliotta G, Saitta S, Polito S, Adile B, Marci R, Calagna G. Is vaginal fractional CO2 laser treatment effective in improving overactive bladder symptoms in post-menopausal patients? Preliminary results. Eur Rev Med Pharmacol Sci. 2016 Jun;20(12):2491-7. PMID 27383297
- [Background] Pitsouni E, Grigoriadis T, Tsiveleka A, Zacharakis D, Salvatore S, Athanasiou S. Microablative fractional CO2-laser therapy and the genitourinary syndrome of menopause: An observational study. Maturitas. 2016 Dec;94:131-136. doi: 10.1016/j.maturitas.2016.09.012. Epub 2016 Sep 16. PMID 27823733
- [Background] Gonzalez Isaza P, Jaguszewska K, Cardona JL, Lukaszuk M. Long-term effect of thermoablative fractional CO2 laser treatment as a novel approach to urinary incontinence management in women with genitourinary syndrome of menopause. Int Urogynecol J. 2018 Feb;29(2):211-215. doi: 10.1007/s00192-017-3352-1. Epub 2017 May 18. PMID 28523400
- [Background] Athanasiou S, Pitsouni E, Antonopoulou S, Zacharakis D, Salvatore S, Falagas ME, Grigoriadis T. The effect of microablative fractional CO2 laser on vaginal flora of postmenopausal women. Climacteric. 2016 Oct;19(5):512-8. doi: 10.1080/13697137.2016.1212006. Epub 2016 Aug 24. PMID 27558459
- [Background] Pitsouni E, Grigoriadis T, Falagas ME, Salvatore S, Athanasiou S. Laser therapy for the genitourinary syndrome of menopause. A systematic review and meta-analysis. Maturitas. 2017 Sep;103:78-88. doi: 10.1016/j.maturitas.2017.06.029. Epub 2017 Jun 27. PMID 28778337
- [Background] Flint R, Cardozo L, Grigoriadis T, Rantell A, Pitsouni E, Athanasiou S. Rationale and design for fractional microablative CO2 laser versus photothermal non-ablative erbium:YAG laser for the management of genitourinary syndrome of menopause: a non-inferiority, single-blind randomized controlled trial. Climacteric. 2019 Jun;22(3):307-311. doi: 10.1080/13697137.2018.1559806. Epub 2019 Jan 24. PMID 30676818
- [Background] Escribano JJ, Gonzalez-Isaza P, Tserotas K, Athanasiou S, Zerbinati N, Leibaschoff G, Salvatore S, Sanchez-Borrego R. In response to the FDA warning about the use of photomedicine in gynecology. Lasers Med Sci. 2019 Sep;34(7):1509-1511. doi: 10.1007/s10103-019-02744-1. Epub 2019 Mar 4. PMID 30830556
- [Background] Lester J, Pahouja G, Andersen B, Lustberg M. Atrophic vaginitis in breast cancer survivors: a difficult survivorship issue. J Pers Med. 2015 Mar 25;5(2):50-66. doi: 10.3390/jpm5020050. PMID 25815692
- [Background] Crandall C, Petersen L, Ganz PA, Greendale GA. Association of breast cancer and its therapy with menopause-related symptoms. Menopause. 2004 Sep-Oct;11(5):519-30. doi: 10.1097/01.gme.0000117061.40493.ab. PMID 15356404
- [Background] Fiorica J. Association of breast cancer and its therapy with menopause-related symptoms. Menopause. 2004 Sep-Oct;11(5):502-4. doi: 10.1097/01.gme.0000131667.98625.42. No abstract available. PMID 15356401
- [Background] Kingsberg SA, Krychman M, Graham S, Bernick B, Mirkin S. The Women's EMPOWER Survey: Identifying Women's Perceptions on Vulvar and Vaginal Atrophy and Its Treatment. J Sex Med. 2017 Mar;14(3):413-424. doi: 10.1016/j.jsxm.2017.01.010. Epub 2017 Feb 12. PMID 28202320
- [Background] Kingsberg SA, Larkin L, Krychman M, Parish SJ, Bernick B, Mirkin S. WISDOM survey: attitudes and behaviors of physicians toward vulvar and vaginal atrophy (VVA) treatment in women including those with breast cancer history. Menopause. 2019 Feb;26(2):124-131. doi: 10.1097/GME.0000000000001194. PMID 30130293
- [Background] Kingsberg SA, Krychman ML. Resistance and barriers to local estrogen therapy in women with atrophic vaginitis. J Sex Med. 2013 Jun;10(6):1567-74. doi: 10.1111/jsm.12120. Epub 2013 Mar 27. PMID 23534861
- [Background] Santen RJ, Stuenkel CA, Davis SR, Pinkerton JV, Gompel A, Lumsden MA. Managing Menopausal Symptoms and Associated Clinical Issues in Breast Cancer Survivors. J Clin Endocrinol Metab. 2017 Oct 1;102(10):3647-3661. doi: 10.1210/jc.2017-01138. PMID 28934376
- [Background] Bygdeman M, Swahn ML. Replens versus dienoestrol cream in the symptomatic treatment of vaginal atrophy in postmenopausal women. Maturitas. 1996 Apr;23(3):259-63. doi: 10.1016/0378-5122(95)00955-8. PMID 8794418
- [Background] Sinha A, Ewies AA. Non-hormonal topical treatment of vulvovaginal atrophy: an up-to-date overview. Climacteric. 2013 Jun;16(3):305-12. doi: 10.3109/13697137.2012.756466. Epub 2013 Jan 8. PMID 23215675
- [Background] Dezzutti CS, Brown ER, Moncla B, Russo J, Cost M, Wang L, Uranker K, Kunjara Na Ayudhya RP, Pryke K, Pickett J, Leblanc MA, Rohan LC. Is wetter better? An evaluation of over-the-counter personal lubricants for safety and anti-HIV-1 activity. PLoS One. 2012;7(11):e48328. doi: 10.1371/journal.pone.0048328. Epub 2012 Nov 7. PMID 23144863
- [Background] Ship JA, McCutcheon JA, Spivakovsky S, Kerr AR. Safety and effectiveness of topical dry mouth products containing olive oil, betaine, and xylitol in reducing xerostomia for polypharmacy-induced dry mouth. J Oral Rehabil. 2007 Oct;34(10):724-32. doi: 10.1111/j.1365-2842.2006.01718.x. PMID 17824884
- [Background] Lopez-Pintor RM, Ramirez L, Serrano J, de Pedro M, Fernandez-Castro M, Casanas E, Hernandez G. Effects of Xerostom(R) products on xerostomia in primary Sjogren's syndrome: A randomized clinical trial. Oral Dis. 2019 Apr;25(3):772-780. doi: 10.1111/odi.13019. Epub 2019 Jan 8. PMID 30561129
- [Background] Martin M, Marin A, Lopez M, Linan O, Alvarenga F, Buchser D, Cerezo L. Products based on olive oil, betaine, and xylitol in the post-radiotherapy xerostomia. Rep Pract Oncol Radiother. 2017 Jan-Feb;22(1):71-76. doi: 10.1016/j.rpor.2016.09.008. Epub 2016 Nov 25. PMID 27920611
- [Background] Villa A, Wolff A, Aframian D, Vissink A, Ekstrom J, Proctor G, McGowan R, Narayana N, Aliko A, Sia YW, Joshi RK, Jensen SB, Kerr AR, Dawes C, Pedersen AM. World Workshop on Oral Medicine VI: a systematic review of medication-induced salivary gland dysfunction: prevalence, diagnosis, and treatment. Clin Oral Investig. 2015 Sep;19(7):1563-80. doi: 10.1007/s00784-015-1488-2. Epub 2015 May 22. PMID 25994331
- [Background] Gil-Montoya JA, Silvestre FJ, Barrios R, Silvestre-Rangil J. Treatment of xerostomia and hyposalivation in the elderly: A systematic review. Med Oral Patol Oral Cir Bucal. 2016 May 1;21(3):e355-66. doi: 10.4317/medoral.20969. PMID 27031061
- [Background] Lopez-Lopez J, Jane Salas E, Chimenos Kustner E. [Prognosis and treatment of dry mouth. Systematic review]. Med Clin (Barc). 2014 Feb 4;142(3):119-24. doi: 10.1016/j.medcli.2013.02.036. Epub 2013 May 31. Spanish. PMID 23726507
- [Background] Valimaa H, Savolainen S, Soukka T, Silvoniemi P, Makela S, Kujari H, Gustafsson JA, Laine M. Estrogen receptor-beta is the predominant estrogen receptor subtype in human oral epithelium and salivary glands. J Endocrinol. 2004 Jan;180(1):55-62. doi: 10.1677/joe.0.1800055. PMID 14709144
- [Background] Leimola-Virtanen R, Salo T, Toikkanen S, Pulkkinen J, Syrjanen S. Expression of estrogen receptor (ER) in oral mucosa and salivary glands. Maturitas. 2000 Aug 31;36(2):131-7. doi: 10.1016/s0378-5122(00)00138-9. PMID 11006500
- [Background] ZISKIN DE, MOULTON R. A comparison of oral and vaginal epithelial smears. J Clin Endocrinol Metab. 1948 Feb;8(2):146-65. doi: 10.1210/jcem-8-2-146. No abstract available. PMID 18907981
- [Background] van der Bijl P, van Eyk AD. Human vaginal mucosa as a model of buccal mucosa for in vitro permeability studies: an overview. Curr Drug Deliv. 2004 Apr;1(2):129-35. doi: 10.2174/1567201043479975. PMID 16305378
- [Background] Morelli L, Zonenenschain D, Del Piano M, Cognein P. Utilization of the intestinal tract as a delivery system for urogenital probiotics. J Clin Gastroenterol. 2004 Jul;38(6 Suppl):S107-10. doi: 10.1097/01.mcg.0000128938.32835.98. PMID 15220672
- [Background] Cribby S, Taylor M, Reid G. Vaginal microbiota and the use of probiotics. Interdiscip Perspect Infect Dis. 2008;2008:256490. doi: 10.1155/2008/256490. Epub 2009 Mar 29. PMID 19343185
- [Background] Mothes AR, Runnebaum M, Runnebaum IB. Ablative dual-phase Erbium:YAG laser treatment of atrophy-related vaginal symptoms in post-menopausal breast cancer survivors omitting hormonal treatment. J Cancer Res Clin Oncol. 2018 May;144(5):955-960. doi: 10.1007/s00432-018-2614-8. Epub 2018 Feb 27. PMID 29487993
- [Background] Becorpi A, Campisciano G, Zanotta N, Tredici Z, Guaschino S, Petraglia F, Pieralli A, Sisti G, De Seta F, Comar M. Fractional CO2 laser for genitourinary syndrome of menopause in breast cancer survivors: clinical, immunological, and microbiological aspects. Lasers Med Sci. 2018 Jul;33(5):1047-1054. doi: 10.1007/s10103-018-2471-3. Epub 2018 Mar 1. PMID 29492713
- [Background] Pieralli A, Fallani MG, Becorpi A, Bianchi C, Corioni S, Longinotti M, Tredici Z, Guaschino S. Fractional CO2 laser for vulvovaginal atrophy (VVA) dyspareunia relief in breast cancer survivors. Arch Gynecol Obstet. 2016 Oct;294(4):841-6. doi: 10.1007/s00404-016-4118-6. Epub 2016 May 12. PMID 27170261
- [Background] Pagano T, De Rosa P, Vallone R, Schettini F, Arpino G, Giuliano M, Lauria R, De Santo I, Conforti A, Gallo A, Nazzaro G, De Placido S, Locci M, De Placido G. Fractional microablative CO2 laser in breast cancer survivors affected by iatrogenic vulvovaginal atrophy after failure of nonestrogenic local treatments: a retrospective study. Menopause. 2018 Jun;25(6):657-662. doi: 10.1097/GME.0000000000001053. PMID 29286986
- [Background] Leone Roberti Maggiore U, Parma M, Candiani M, Salvatore S. Microablative Fractional CO2 Laser for Vulvovaginal Atrophy in Women With a History of Breast Cancer. J Minim Invasive Gynecol. 2015 Nov-Dec;22(6S):S100. doi: 10.1016/j.jmig.2015.08.269. Epub 2015 Oct 15. No abstract available. PMID 27678561
- [Background] Jha S, Wyld L, Krishnaswamy PH. The Impact of Vaginal Laser Treatment for Genitourinary Syndrome of Menopause in Breast Cancer Survivors: A Systematic Review and Meta-analysis. Clin Breast Cancer. 2019 Aug;19(4):e556-e562. doi: 10.1016/j.clbc.2019.04.007. Epub 2019 Apr 19. PMID 31227415
- [Background] Gambacciani M, Levancini M, Cervigni M. Vaginal erbium laser: the second-generation thermotherapy for the genitourinary syndrome of menopause. Climacteric. 2015 Oct;18(5):757-63. doi: 10.3109/13697137.2015.1045485. PMID 26029987
- [Background] Robinson D, Flint R, Veit-Rubin N, Araklitis G, Cardozo L. Is there enough evidence to justify the use of laser and other thermal therapies in female lower urinary tract dysfunction? Report from the ICI-RS 2019. Neurourol Urodyn. 2020 Jul;39 Suppl 3:S140-S147. doi: 10.1002/nau.24298. Epub 2020 Feb 10. PMID 32040871
- [Background] Alvisi S, Baldassarre M, Martelli V, Gava G, Seracchioli R, Meriggiola MC. Effects of ospemifene on vaginal epithelium of post-menopausal women. Gynecol Endocrinol. 2017 Dec;33(12):946-950. doi: 10.1080/09513590.2017.1332589. Epub 2017 May 31. PMID 28562130
- [Background] Alvisi S, Baldassarre M, Gava G, Mancini I, Gagliardi M, Seracchioli R, Meriggiola MC. Structure of Epithelial and Stromal Compartments of Vulvar and Vaginal Tissue From Women With Vulvo-Vaginal Atrophy Taking Ospemifene. J Sex Med. 2018 Dec;15(12):1776-1784. doi: 10.1016/j.jsxm.2018.10.009. Epub 2018 Nov 13. PMID 30446472
- See also: Spanish Agency for Medicines and Health Products. SmPC Blissel 50 micrograms/gram vaginal gel — http://cima.aemps.es/cima/pdfs/es/ft/72726/FichaTecnica_72726.html.pdf
- See also: EUROPEAN MEDICINES AGENCY. Data sheet Prasterone 6.5 milligrams — http://www.ema.europa.eu/en/documents/product-information/intrarosa-epar-product-information_es.pdf
- See also: EUROPEAN MEDICINES AGENCY. Technical Sheet Ospemifene 60 mg — http://www.ema.europa.eu/en/documents/product-information/senshio-epar-product-information_es.pdf